CLINICAL TRIAL: NCT04655001
Title: MORPH II: Revisiting A Mobile Intervention to Reduce Pain and Improve Health (MORPH)
Brief Title: Revisiting A Mobile Intervention to Reduce Pain and Improve Health
Acronym: MORPH-II
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Principal Investigator, Jason Fanning, Assistant Professor, Wake Forest University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00023965
Record Dates: First submitted 2020-12-03; First posted 2020-12-04 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Pain; Obesity; Sedentary Behavior
Keywords: Telehealth; Aging; mHealth; Wearable
MeSH Terms: conditions — Pain; Obesity; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to a 24-week intervention or a no-contact control
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MORPH (Experimental): Participants engage in 12 weeks of group and 1-on-1 coaching meant to promote physical activity throughout the day and caloric restriction. Participants engage with a custom smartphone application, use a smart scale and physical activity monitor, and meet using video conference software. At the end of 12 weeks, participants are provided with tools to continue meeting virtually on their own if desired, and will be followed for an additional 12-week maintenance phase.
  Interventions: Behavioral: MORPH
- Control (No Intervention): This condition receives the wearable activity monitor and simply asked to use it and continue in their daily lives for 24 weeks.

INTERVENTIONS:
Behavioral: MORPH — A 12-week movement and caloric restriction intervention meant to reduce pain and body weight.
  Arms: MORPH

SUMMARY:
Chronic pain is a pervasive and costly health condition among older adults that is associated with wide-ranging adverse health outcomes including falls, declining mobility, and increasing functional disability. Obesity exacerbates many of these health issues, contributing to a higher frequency of intractable pain episodes, increased pain severity, multi-site pain, and the use of stronger opioid medications compared to normal weight individuals with chronic pain. In addition, older adults who suffer from chronic pain are significantly more sedentary than those without chronic pain. Despite evidence relating increased sedentary behavior to pain, non-pharmacological treatments have largely focused on structured moderate-to-vigorous physical activity (MVPA) by way of conventional forms of exercise.

Recent evidence from an intervention designed to decreased sedentary behavior (SB) demonstrated the approach is effective in preventing weight regain following weight loss. A subsequent study-a mobile intervention to reduce pain and improve health (MORPH: Wake Forest Baptist Health institutional review board [IRB] 00046364)-demonstrated that a primarily home-delivered intervention (9 of 12 delivered in home; 3 of 12 delivered in a research center) supported by technology can produce significant weight loss, reductions in sedentary time, increases in daily steps, less pain intensity, and better physical function compared with a waitlist control. MORPH included a focus on dietary weight loss plus movement across the day through a combination of group telecoaching and a custom mobile health (mHealth) application, but results indicated that participants did not internalize the day-long movement intervention. Instead, they appeared to achieve a greater number of steps through conventional walking exercise, allowing for high levels of sitting, stiffness, and pain.

MORPH concluded with a two-group randomized controlled pilot trial (RCT) in obese (BMI=30-45 kg/m2), low-active, older (55-85 years) adults with chronic pain who were randomized to either 12-weeks of active intervention or a wait-list control. This study represents an extension of MORPH-hereafter MORPH II-with the intention of immediately addressing limitations in the original MORPH study. Participants will be randomize 30 older, low-active, obese adults to the active intervention or to a standard control for 12 weeks. To build upon the last phase of MORPH, the research team will deliver this intervention fully remotely, providing cellular data-equipped tablet computers to protect participant safety and reduce technical issues that may arise due to lack of face-to-face orientation appointments. Given the current COVID-19 climate, the investigators have chosen to deliver the entire intervention remotely. The investigators are implementing intensive individual coaching throughout the program and greater emphasis on frequent movement to drive better uptake of a day-long movement program and will transition participants to a 12-week no-contact follow-up to observe whether behavior change sustains following completion of the focused intervention.

This study is couched within a contemporary engineering-inspired design framework-the multiphase optimization strategy (MOST)-which emphasizes rapid identification of successful intervention components and the removal or redesign of components that are either ineffective or perceived as a nuisance. To this end, the study team will carry momentum from MORPH into MORPH II wherein the team will assess the impact of a fully remote MORPH intervention with the addition of high-contact coaching on pain ratings, physical function, levels of physical activity and sedentary behavior, and body weight. This is particularly timely given limited access to center-based resources for many during the COVID-19 pandemic, and especially those who are high-risk, including older adults with chronic pain.

Aims and Hypotheses Specific Aim 1: To conduct a pilot RCT to provide initial evidence for the effect size associated with the proposed intervention on pain, sitting time, and daily steps. Investigators will also explore the impact of this program on social connection (i.e., relatedness) and physical function.

Hypothesis 1: It is expected that the provision of the in-home application to contribute to clinically meaningful improvements in pain ratings and steps and a reduction in daily sedentary time compared to the control condition.

Specific Aim 2: To examine whether a socially mediated, home-delivered health intervention produces lasting behavior change over a 12-week no-contact period.

Hypothesis 2: It is expected that levels of physical activity at week 24 will remain meaningfully improved over baseline in the intervention condition relative to the control.

ELIGIBILITY:
Inclusion Criteria:

* Age 55-85 years;
* Corrected (based on phone self-reported height and weight) BMI=30-45 kg/m2;
* Has data coverage in the home;
* Weight stable-reporting no loss or gain (±5%) in past 6 months;
* Willing to provide informed consent;
* Agree to all study procedures and assessments;
* Owns an Android or Apple smartphone;
* Self-reported pain in 2 or more of the following sites on most days for the previous 3 months: back, neck, shoulders, hips and/or knees

Exclusion Criteria:

* Dependent on cane or walker to walk a short distance; >1 fall (injurious or non-injurious) in past year (does not include falls where participant was pushed/pulled by another object and was not injured)
* Vision insufficient to read a smartphone screen, unable to read
* Participation in regular resistance training and/or > 20 mins on 2+ d/w of aerobic exercise in past 6 months
* No contraindication to exercise
* TICS-M score ≤ 31
* Uncontrolled hypertension (>160/90 mmHg);
* Current or recent past (within 1 year) severe symptomatic heart disease, uncontrolled angina, stroke, osteoporosis, chronic respiratory disease requiring oxygen, neurological or hematological disease; cancer requiring treatment in past yr, except non-melanoma skin cancers
* Regular use of: growth hormones, oral steroids, or prescription osteoporosis medications
* Current participation in other research study targeting pain, physical activity, or weight loss.
* Previous participation in MORPH I- phase 1 or 2
* Joint replacement or orthopedic surgery within previous 6 months or planning to have orthopedic surgery in the next 6 months

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Baseline to week 12
  PROMIS (Patient-Reported Outcomes Measurement Information System) 3-item pain intensity scale. Final scores represent t-scores (mean of 50, standard deviation of 10) where greater scores represent greater pain intensity relative to a nationally representative sample.
Pain Interference | Baseline to week 12
  PROMIS (Patient-Reported Outcomes Measurement Information System) 8-item pain interference scale. Final scores represent t-scores (mean of 50, standard deviation of 10) where greater scores represent greater pain interference relative to a nationally representative sample.
Steps | Baseline to week 12
  Daily steps as recorded by the ActivPAL accelerometer.
Sedentary time | Baseline to week 12
  Daily minutes spent sedentary as recorded by the ActivPAL accelerometer.

SECONDARY OUTCOMES:
Steps | Baseline to week 24
  Daily steps at 24 weeks as recorded by the ActivPAL accelerometer.

OTHER OUTCOMES:
Physical Function | Baseline to week 12
  Physical function as assessed by the short physical performance battery. Scores are on a scale of 0 - 12 with higher scores representing better physical functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Fanning, PhD, Principal Investigator — Wake Forest University
Locations (1):
- Wake Forest University, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fanning J, Brooks AK, Ip E, Nicklas BJ, Rejeski WJ. A Mobile Health Intervention to Reduce Pain and Improve Health (MORPH) in Older Adults With Obesity: Protocol for the MORPH Trial. JMIR Res Protoc. 2018 May 14;7(5):e128. doi: 10.2196/resprot.9712. PMID 29759957
- [Derived] Fanning J, Brooks AK, Hsieh KL, Kershner K, Furlipa J, Nicklas BJ, Rejeski WJ. Building on Lessons Learned in a Mobile Intervention to Reduce Pain and Improve Health (MORPH): Protocol for the MORPH-II Trial. JMIR Res Protoc. 2021 Jul 19;10(7):e29013. doi: 10.2196/29013. PMID 34279241